CLINICAL TRIAL: NCT01139944
Title: Epigenetic Changes as Prognostic Markers in Patients With Early Stage Non-Small Cell Lung Cancer
Brief Title: Biomarkers in Tissue and Blood Samples From Patients With Early-Stage Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z4102; ACOSOG-Z4102; CDR0000671680 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — DNA Methylation; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Archived tumor and intrathoracic lymph node tissue samples are analyzed for aberrant DNA methylation (p16/CDKN2A, DAP kinase, H-cadherin, APC, and RASSF1A) by methylation-specific PCR. Analyses are then compared with the preliminary data from the Johns Hopkins institutional study.
  Interventions: Genetic: DNA methylation analysis; Genetic: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue and blood samples from patients with early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate aberrant methylation patterns in tissue and serum samples from patients with early-stage non-small cell lung cancer (NSCLC) to validate the Johns Hopkins single institutional study.
* Attempt to define subgroups of patients at greater risk for recurrent or metastatic disease who may benefit from more aggressive adjuvant therapeutic regimens.
* Develop prognostic indicators for disease-specific and overall survival.
* Define new potential molecular targets for therapy.

OUTLINE: Archived tumor and intrathoracic lymph node tissue samples are analyzed for aberrant DNA methylation (p16/CDKN2A, DAP kinase, H-cadherin, APC, and RASSF1A) by methylation-specific PCR. Analyses are then compared with the preliminary data from the Johns Hopkins institutional study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of early-stage non-small cell lung cancer

  * T1 or T2, N0 disease
  * Had a lobectomy or greater resection with negative surgical margins (R0 resection)
* Available tumor and lymph node specimens from patients enrolled on ACOSOG-Z0040 and ACOSOG-Z0030 trials

  * Node-negative with recurrent disease within 3 years (cases)
  * Node-negative patients without recurrent disease (controls)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with early stage non-small cell lung cancer and previously enrolled on ACOSOG-Z0040 and Z0030.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
disease specific survival | Up to 10 years
overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm V. Brock, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins